CLINICAL TRIAL: NCT01023412
Title: Effect of 3 Day Pre-operative Immunonutrition Regimen on Clinical Outcome in Well-nourished Patients With Gastrointestinal Cancer Undergoing Surgery , a Randomised Double-blind Controlled Trial
Brief Title: Effects of 3 Day Preoperative Immunonutrition in Well-nourished Patients With Gastrointestinal (GI) Cancer Undergoing Surgery
Acronym: IPOD-3
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: interim review of the data indicated that the hypothesis put forth on the efficacy of a 3 day regimen was not met.
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SC-IRTD-01-05-CH
Record Dates: First submitted 2009-11-16; First posted 2009-12-02 (Estimated); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Gastrointestinal Cancer
Keywords: Immunonutrition; cancer; GI cancer surgery
MeSH Terms: conditions — Gastrointestinal Neoplasms; Neoplasms | interventions — Immunonutrition Diet

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutritional product (Active Comparator): Oral nutritional supplement containing immuno nutrients
  Interventions: Dietary Supplement: Immunonutrition
- Isocaloric control (Placebo Comparator): Isocaloric and isonitrogenous control without immuno nutrients
  Interventions: Dietary Supplement: Immunonutrition

INTERVENTIONS:
Dietary Supplement: Immunonutrition — Oral Nutritional Supplement containing the amino acid arginine, omega-3 fatty acids, and nucleotides (RNA).

SUMMARY:
Major surgery is still associated with a high rate of postoperative morbidity despite improved techniques in surgical management. Surgery-induced alterations of the immune system are well described and may play a role in the genesis of postoperative complications. It has been shown by several large scale clinical trials, that the use of immunonutrition in postoperative cancer surgery, trauma and critically ill patients resulted in an improved immunocompetence and/or reduced postoperatively infectious morbidity and/or length of hospital stay.The pre-operative regimen was between 5 to 7 days of treatment. The aim of this trial is to evaluate if a shorter administration of 3 days pre-operatively would be beneficial as well.

ELIGIBILITY:
Inclusion Criteria:

* Patients with GI cancer (stomach, pancreas, small and large bowel and rectum) histologically proven
* Well nourished patients as defined by a total score of <3 on the nutritional screening tool NRS-2002 (46) (Appendix III)
* Patients who are >= 18 years of age;
* Patients who have signed a written Informed Consent (Appendix I) prior to admission to the study;
* Patients who have an ECOG performance status of 0, 1 or 2 (Appendix II).
* Patients able to orally consume 750 mL or more of liquid a day prior to surgery

Exclusion Criteria:

* Patients who have co-morbid conditions, uncontrolled metabolic conditions or psychiatric conditions that might make tolerance or evaluation of the feeding formula difficult;
* Patients who are pregnant;
* Patients with cardiac failure as defined by the Goldman classification class>3
* Patients with respiratory failure (FEV<0.8l/sec)
* Patients with renal failure (Cr >= 3mg/dl or dialysis patients)
* Patients with hepatic dysfunction (Child >A)
* Patients suffering from an intestinal obstruction or ileum
* Patients with an Hb level of <=8 g/dL experiencing gastrointestinal hemorrhaging
* Patients with HIV, HCV, HBV
* Patients requiring immunosuppression treatments
* Patients undergoing emergency surgery
* Other patients determined by a study investigator to be inappropriate for enrolment in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2006-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Rate of post-operative complications | On the day of discharge from hospital

SECONDARY OUTCOMES:
Incidence of non-infectious complications | On the day of discharge from hospital
Length of hospital stay | On the day of discharge from hospital
Nutritional status evaluation | On the day of discharge from hospital
Rate of post-operative infectious complications | On the day of discharge from hospital

CONTACTS AND LOCATIONS:
Locations (6):
- Switzerland (6):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden, Baden
  - Lindenhof-Spital, Bern
  - Kantonsspital Liestal, Liestal
  - Kantonsspital St.Gallen, Sankt Gallen
  - Kantonsspital Schaffausen, Schaffhausen